CLINICAL TRIAL: NCT03181061
Title: Determinants of Success, Characterizing the Facilitators of Integrated Abortion Provision
Acronym: FAB
Status: Withdrawn | Type: Observational
Why Stopped: PI confirmed that this is not a clinical trial and was inadvertently entered in the system
Sponsor: University of New Mexico (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Other Study IDs: 17-124
Record Dates: First submitted 2017-06-05; First posted 2017-06-08 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy Termination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Semi-structured interviews — Providers will participate in a semi-structured interview using an interview guide that addresses 4 domains of interest including: (1) initiation of abortion services, (2) barriers to abortion provision, (3) facilitators of abortion provision and (4) acquired expertise and coaching for success.

SUMMARY:
This national, qualitative study of physicians who provide abortion care aims to better understand the facilitators of abortion provision among generalist clinicians in OB-GYN and Family Medicine.

DETAILED DESCRIPTION:
This is a nationwide qualitative study of 20 to 40 physicians who provide abortion services as part of their scope of practice. Providers will participate in a semi-structured interview using an interview guide that addresses 4 domains of interest including: (1) initiation of abortion services, (2) barriers to abortion provision, (3) facilitators of abortion provision and (4) acquired expertise and coaching for success.

ELIGIBILITY:
Inclusion Criteria:

* Practicing obstetrician-gynecologists and family medicine physicians who currently provide or in the past have provided abortion services (medication abortions, surgical abortions and/or induction abortions) as part of their clinical practice will be eligible for study participation.
* All providers who meet these criteria will be eligible regardless of providers' gestational age cutoff, abortion indication limitations and/or restrictions, or number of abortions provided.

Exclusion Criteria:

* Physicians who work solely at a designated abortion facility, e.g., Planned Parenthood, without an alternate practice site, or who provide only abortions, are not eligible for study participation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Providers of Abortion Care
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Integration of Abortion Care | April 2017-February 2018
  To qualitatively interview obstetrician/gynecologists and Family Medicine physicians who have successfully integrated abortion care into their practice scope and to explore their experiences with abortion provision.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hofler, MD, MBA, MPH, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No